CLINICAL TRIAL: NCT02684552
Title: Physiotherapist in Charge of the Study
Brief Title: Non Invasive Ventilation During Physical Training in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Cecilia Rodriguez, Physiotherapist, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Noninvasive Ventilation; Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non invasive ventilation (Experimental): Patients perform physical test with non invasive ventilation
  Interventions: Device: Non invasive ventilation
- Oxygen (Active Comparator): Patients perform physical test with oxygen with mask
  Interventions: Device: Oxygen

INTERVENTIONS:
Device: Non invasive ventilation — Training on treadmill with Non invasive ventilation
  Arms: Non invasive ventilation
Device: Oxygen — Training on treadmill with oxygen
  Arms: Oxygen

SUMMARY:
Patients with cystic fibrosis older than 18 years will performance a Bruce test with non invasive ventilation (once) after 30 minutes they perform the same test with oxygen supplementation.

Measurements: Transcutaneous level off carbon dioxide, saturation, puls and dyspnea scale.

DETAILED DESCRIPTION:
measurements before and after the test: transcutaneous level off carbon dioxide, saturation, respiratory rate, dyspnea scale.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Cystic Fibrosis at Stockholm Cystic Fibrosis center
* > 18 years of age
* Forced expiratory volume in one second (FEV1) between 20 and 69% of predicted value
* Developed alveolar hypoventilation at the physical performance test
* Use oxygen supplementation during aerobic training

Exclusion Criteria:

* Symptomatic upper airway infection characterized by fever less than 1 month before entering the study
* Cognitive dysfunction
* Cardio-respiratory instability
* Infection with Burkholderia cepacia complex
* Gastroesophageal reflux
* History of pneumothorax
* Massive hemoptysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Transcutaneous level carbon dioxide | 10 min measurement
  Physiological parameter

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cecilia Rodriguez Hortal, MSC, Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Cecilia Rodriguez, Stockholm, Stockholm County
  - Maria Cecilia Rodriguez Hortal, Stockholm

IPD SHARING:
Plan to Share IPD: No